CLINICAL TRIAL: NCT05994677
Title: Psoriasis and Non Alcoholic Steatohepatitis: Is There a Shared Inflammatory Network ?
Acronym: PANASH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Mohamed Hussein, Resident doctor, Assiut University
Other Study IDs: AssiutUFMGIT
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Nash
Keywords: NASH; Psoriasis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is to assess frequency of NASH in Psoriatic patient and to measure the level of proinflammatory cytokines including TNFα, interleukin (IL)-6 and IL-17 and anti-inflammatory cytokines including IL10, IL35 by ELISA.

DETAILED DESCRIPTION:
• Psoriasis is a chronic proliferative and inflammatory condition of the skin. It is characterized by erythematous plaques covered with silvery scales, particularly over the extensor surfaces, scalp, and lumbosacral region.

The disorder can also affect the joints and eyes. Psoriasis has no cure and the disease waxes and wanes with flareups. There are several subtypes of psoriasis but the plaque type is the most common and presents on the trunk, extremities, and scalp.

Psoriasis has a prevalence ranging from 0.2% to 4.8%.

In parallel, nonalcoholic fatty liver disease (NAFLD) is the most frequent liver disease worldwide, affecting an estimated 30% of the adult population in developed countries.

NAFLD and the metabolic syndrome are mutually and bi-directionally associated, as these two pathologic condition share insulin resistance as a common pathophysiological mechanism.

NAFLD encompasses a spectrum of pathologic conditions ranging from simple steatosis to nonalcoholic steatohepatitis((NASH) featuring steatosis associated with inflammatory changes, hepatocellular ballooning and pericellular fibrosis), to advanced fibrosis and cirrhosis. NAFLD is projected to become the most common indication for liver transplantation in the United States by 2030 .

Over the last few years, multiple studies have demonstrated that psoriasis is associated with NAFLD. The majority reported a prevalence of around 50 % (range 14.4 % to 65.5 %) for NAFLD in psoriatic patients.

The contribution of IL-17 to the pathogenesis of both psoriasis and NAFLD is intriguing. Th17 cells can be detected in fat tissue and IL-17 itself regulates glucose metabolism and adipogenesis. Likewise, IL-17(A)-secreting Th17 cells may promote the progression from simple steatosis to steatohepatitis [10] Therefore, both psoriasis and NAFLD pathogenesis seem to be linked to the joint proinflammatory Th17 axis (and other cytokines such as TNFα and IL-6).

ELIGIBILITY:
Inclusion Criteria:

* Any naive psoriatic patient above 18 years old.

Exclusion Criteria:

* Any psoriatic patient who received treatment for psoriasis.
* Diabetic patients.
* Patients under 18 years old.
* Patient's refusal.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Psoriatic patients above 18 years not diabetic and not receiving treatment for psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Main | Baseline
  To find out if there is a shared inflammatory network between psoriasis and Non Alcoholic Steatohepatitis or not.

SECONDARY OUTCOMES:
subsidiary | Baseline
  Incidence of Non Alcoholic Steatohepatitis in psoriatic patients.

IPD SHARING:
Plan to Share IPD: No